CLINICAL TRIAL: NCT02060513
Title: Rapid Microbiological Diagnostics for MDRO Quantitative Identification and Resistance Phenotyping to Guide Antibiotic Selection in Wounded Warriors and Veterans
Brief Title: Study of Accuracy of New Diagnostic Technology to Determine Guide Rapid Antibiotic Treatment for Serious Infections
Acronym: RAMPED
Status: Completed | Type: Observational
Sponsor: Connie Price (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Accelerate Diagnostics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Connie Price, Professor, Denver Health and Hospital Authority
Organization: Denver Health and Hospital Authority (Other)
Other Study IDs: 12-1580; W81XWH-12-2-0085 (Other: Department of Defense)
Record Dates: First submitted 2014-02-03; First posted 2014-02-12 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2016-12

CONDITIONS: Infection; Skin and Subcutaneous Tissue Bacterial Infections; Healthcare-associated Infection; Infection Due to Resistant Bacteria
Keywords: Wounded warriors; Battlefield infection; Acinetobacter; ESBL; MRSA; KPC
MeSH Terms: conditions — Infections; Cross Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Isolates of intresting bacteria
Oversight: Data Monitoring Committee: No

SUMMARY:
Military service members and the U.S. veteran population face a growing and serious health threat: widespread antibiotic resistance resulting from resistant bacteria and a dwindling pipe-line of sufficiently potent antibiotics. Infections with antibiotic resistant bacteria are increasing significantly. They cause major complications and mortality, and drive up healthcare costs. Powerful but non-targeted antibiotics, while in widespread use, can actually pressure bacteria to develop resistance.

DETAILED DESCRIPTION:
Current methods for diagnosing infections typically require 2-3 days to produce results that can guide antibiotic choice. That is frequently too delayed to help clinicians make good treatment decisions. This also results in inappropriate or over-treatment with non-targeted antibiotics that are started while awaiting lab results. More rapid technologies that can accurately diagnose the specific cause of an infection could guide early, targeted antibiotic treatment. This would result in more effective early treatment of infection, decrease unnecessary exposure to excess antibiotics, and could slow the development of antibiotic resistance. By diagnosing infections earlier, we expect to reduce the complications and mortality of combat-related infections in Wounded Warriors and Military Veterans.

We propose a new ultra-rapid technology (called MADM) that uses a digital microscope to detect bacteria growing directly from a patient's specimen, rather than waiting for growth in lab cultures. The innovative new method supports identification of the infecting bacteria within 2 hours of receiving a specimen. The technology also shows the effect of selected antibiotics on the bacteria including multidrug resistant bacteria so that doctors know within 6 hours from specimen collection which antibiotic kills the bacteria.

This study involves collection of any excess volume of microbiology specimens after it has been determined sufficient sample is available for clinical care. All microbiological samples and results are being obtained for solely non-research purposes as part of usual care; only leftover/discarded materials from clinical or research procedures already performed will be used for this study. Samples will be tested in tandem with usual care on the new technology to test the accuracy and speed. Results obtained from the new technology will not be used in patient care or to make treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Microbiology culture (respiratory, blood or tissue/skin) ordered during regular clinical care.

Exclusion Criteria:

* Insufficient sample volume available after clinical test completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with a suspected infection.
Sampling Method: Non-Probability Sample
Enrollment: 2298 (Actual)
Dates: Start 2013-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The proportion of concordant, accurately phenotyped positive isolates assayed by MADM versus conventional culture based microbiology as comparator. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Connie S Price, MD, Principal Investigator — Denver Health Medical Center; Ivor S Douglas, MD, Principal Investigator — Denver Health Medical Center
Locations (3):
- United States (3):
  - Denver Health Medical Center, Denver, Colorado
  - Denver Veterans Affairs Eastern Colorado Health Care System, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia